CLINICAL TRIAL: NCT00516919
Title: Controlled Trial of Orlistat With Behavioral Weight Loss Therapy for Obesity and Binge Eating in Monolingual Hispanic Persons
Brief Title: Study of Behavioral Weight Loss Therapy for Obesity and Binge Eating in Monolingual Hispanic Persons
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Donaghue Medical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0608001753
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Results first posted 2013-02-07 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Obesity; Binge Eating
Keywords: Obesity; Binge Eating; Monolingual Hispanic Persons; Orlistat; Behavioral Weight Loss Treatment
MeSH Terms: conditions — Obesity; Bulimia | interventions — Orlistat; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Xenical + behavioral intervention
  Interventions: Drug: Xenical + behavioral intervention
- 2 (Active Comparator): Placebo + behavioral intervention
  Interventions: Behavioral: Behavioral intervention + placebo

INTERVENTIONS:
Drug: Xenical + behavioral intervention — 120 mg TID; Behavioral weight loss in Spanish
  Other Names: Xenical
  Arms: 1
Behavioral: Behavioral intervention + placebo — Behavioral weight loss treatment in Spanish Placebo TID
  Arms: 2

SUMMARY:
This is a research study designed to examine the effectiveness of an obesity medication (orlistat) given in addition to behavioral weight loss therapy. Participants will be obese monolingual (Spanish-speaking only) men and women.

ELIGIBILITY:
Inclusion Criteria:

* Monolingual Spanish Speaking
* Obese (BMI >= 30)

Exclusion Criteria:

* Pregnancy
* Current cardiac disease
* Serious neurologic illnesses

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2007-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Grilo, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Hispanic Clinic of the Connecticut Mental Health Center, New Haven, Connecticut
  - Yale Department of Psychiatry, New Haven, Connecticut

REFERENCES:
- [Derived] Grilo CM, Kerrigan SG, Lydecker JA, White MA. Physical activity changes during behavioral weight loss treatment by Latinx patients with obesity with and without binge eating disorder. Obesity (Silver Spring). 2021 Dec;29(12):2026-2034. doi: 10.1002/oby.23278. Epub 2021 Sep 28. PMID 34582624
- [Derived] Grilo CM, White MA. Orlistat with behavioral weight loss for obesity with versus without binge eating disorder: randomized placebo-controlled trial at a community mental health center serving educationally and economically disadvantaged Latino/as. Behav Res Ther. 2013 Mar;51(3):167-75. doi: 10.1016/j.brat.2013.01.002. Epub 2013 Jan 18. PMID 23376451

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled participants from August 2007 through October 2009. Participants were a consecutive series of 79 monolingual (Spanish-speaking-only) obese Latino/as recruited from clinical teams and referrals at a community mental health center serving economically disadvantaged persons with mental health needs.
Groups:
- Xenical + Behavioral Intervention: Drug: Xenical + Behavioral: behavioral intervention
  Xenical + behavioral intervention : 120 mg three times a day; Behavioral weight loss in Spanish
- Placebo + Behavioral Intervention: Drug: Placebo + Behavioral: behavioral intervention
  Behavioral intervention + placebo : Behavioral weight loss treatment in Spanish Placebo three times a day
Period: Overall Study
Arm/Group | Xenical + Behavioral Intervention | Placebo + Behavioral Intervention
Started | 40 | 39
Completed | 30 | 32
Not Completed | 10 | 7

BASELINE CHARACTERISTICS:
Arm/Group | Total Enrollment
Number analyzed (Participants) | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 79
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 79

OUTCOME MEASURES:

1. Primary Outcome: Participant BMI
Description: Body Mass Index (BMI)
Time Frame: 4 months and 6 month follow-up
Population: Data for all randomized participants were included. In the event of dropout or missing data, baseline values were used.
Measure: Mean (Standard Deviation); unit: kg/m^2
Groups:
- Drug: Xenical + Behavioral: Behavioral Intervention: Xenical + behavioral intervention
  Xenical + behavioral intervention : 120 mg three times a day; Behavioral weight loss in Spanish
- Drug: Placebo + Behavioral: Behavioral Intervention: Placebo + behavioral intervention
  Behavioral intervention + placebo three times a day: Behavioral weight loss treatment in Spanish Placebo TID
Arm/Group | Drug: Xenical + Behavioral: Behavioral Intervention | Drug: Placebo + Behavioral: Behavioral Intervention
Number analyzed (Participants) | 40 | 39
kg/m^2
  Post-treatment (4 months) | 36.0 (5.9) | 36.4 (4.7)
  6 month follow up | 36.3 (4.9) | 36.8 (4.7)
Statistical Analysis 1: Comparison: Drug: Xenical + Behavioral: Behavioral Intervention vs Drug: Placebo + Behavioral: Behavioral Intervention; Test for group differences in BMI at post-treatment, controlling for baseline BMI; Test type: Superiority or Other; p = 0.51, ANCOVA; Covariate = Baseline (pre-treatment) BMI; Degrees of freedom = (1, 76); F statistic = 0.45
Statistical Analysis 2: Comparison: Drug: Xenical + Behavioral: Behavioral Intervention vs Drug: Placebo + Behavioral: Behavioral Intervention; Test for group differences in BMI at 6-month follow-up, controlling for baseline BMI; Test type: Superiority or Other; p = 0.41, ANCOVA; Covariate = Baseline (pre-treatment) BMI; Degrees of freedom = (1, 76); F statistic = 0.69

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the trial (through 4 months of active treatment).
Description: Overall frequency of reported side effects was only slightly higher for Xenical than for placebo, although reports of minor gastrointestinal events known to be due to Xenical's mechanism of action were higher for the Xenical condition. Nearly all events occurred early in treatment, were generally mild, and resolved spontaneously.
Groups:
- Drug: Placebo + Behaviora: Behavioral Intervention: Placebo + behavioral intervention
  Behavioral intervention + placebo three times a day: Behavioral weight loss treatment in Spanish Placebo TID
Arm/Group | Drug: Xenical + Behavioral: Behavioral Intervention | Drug: Placebo + Behaviora: Behavioral Intervention
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 0/40 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No